CLINICAL TRIAL: NCT05764850
Title: Mechanisms of Type 1 Diabetes Endophenotypes, by Cluster Analysis
Brief Title: Mechanisms of Type 1 Diabetes Endophenotypes
Acronym: METYDIA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Pediatric Clinical Research Platform (Other)
Collaborators: University Hospital, Geneva (Other); University of Geneva, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-02119
Record Dates: First submitted 2023-02-16; First posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-02

CONDITIONS: Type 1 Diabetes Mellitus; Genetic Predisposition to Disease
Keywords: Type 1 diabetes mellitus; Children; Adolescent; Young adult; Genetic; Transcriptomic; Metabolomic; Lipidomic; Genetic risk score
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Genetic Predisposition to Disease; Genetic Risk Score

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: 100 patients followed in pediatric diabetology at the university hospital of Geneva: a cohort
  Interventions: Genetic: Genome sequencing
- Control: 50 control patients
  Interventions: Genetic: Genome sequencing

INTERVENTIONS:
Genetic: Genome sequencing — 100 extensively phenotyped pediatric and young adult patients for genotyping, metabolomic and lipidomic analyses. Polygenic risk scores for type 1 diabetes and cardiovascular disease will be performed.
  For patients older than 6 years who agree to do a second visit (optional), a Mixed Meal Tolerance Test (MMTT: the gold standard for assessing beta cell function) will be done as well as transcriptomic analysis.
  Other Names: Lipidomic; Metabolomic; Transcriptomic; Mixed meal tolerance test

SUMMARY:
The goal of this observational study consists of performing cluster analysis to decipher underlying disease mechanisms of type 1 diabetes in children and young adults.

To this end, we will combine clinical, laboratory, genetic, transcriptomic, and metabolomic datasets of an extensively phenotyped cohort of children and young adults with type 1 diabetes. We will also assess the risk for cardiovascular diseases in this most vulnerable diabetes cohort.

ELIGIBILITY:
Inclusion Criteria (Type 1 Diabetic patients):

* Informed consent as documented by signature
* Patient's age: between 0 and 25 years old.
* Children, adolescents, and young adult patients followed in diabetology.

Exclusion Criteria (Type 1 Diabetic patients):

* No exclusion criteria

Inclusion Criteria (Controls):

* Informed consent as documented by signature
* Patient's age: 25 less than 6 years of age and 25 between 6 and 25 years old.
* Healthy patient

Exclusion Criteria (Controls):

* Patient receiving treatment affecting metabolic control (ex: systemic corticoids, beta blocker, immunotherapy etc.)
* Concomitant disease that may affect the analysis of the results (ex: cancer, active autoimmune disease requiring treatment)

Ages: 0 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children, adolescents, and young adults followed at the pediatric diabetology unit of the University Hospital of Geneva.
  Controls Children, adolescents, and young adults coming for a routine blood sample at University Hospital of Geneva
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Cluster analysis to decipher underlying mechanisms of type 1 diabetes | blood sampling and analyses
  We will combine clinical, laboratory, genetic, transcriptomic, and metabolomic datasets of an extensively phenotyped cohort of type 1 diabetes patients (Children and young adults).
  We will create clinical and genetic correlates with the following clinical parameters: Age at diabetes onset (years), disease duration (years), BMI (kg/m2), diabetes autoantibodies, C-peptide level (pmol/l) and decline over time, HbA1c (%), insulin dose (U/kg/d), ketoacidosis at disease onset (y/n), lipid levels (Total cholesterol, triglycerides, HLD, LDL, Lipoprotein(a)), macro- and microvascular complications, ethnicity, family history for diabetes, associated autoimmune diseases (e.g., autoimmune thyroiditis or celiac disease) and mixed meal tolerance test.

CONTACTS AND LOCATIONS:
Overall Officials: Valerie VS Schwitzgebel, MD, Principal Investigator — University Hospital of Geneva / University of Geneva
Locations (1):
- University Hospital of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No